CLINICAL TRIAL: NCT03636490
Title: Psychological Stress, and Circadian Patterns of Sodium Excretion and Blood Pressure
Brief Title: Stress, Salt Excretion, and Nighttime Blood Pressure
Acronym: SABRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Daichi Shimbo, Professor of Medicine, Dept of Med, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAS0154; 1R01HL137818-01A1 (NIH)
Record Dates: First submitted 2018-08-09; First posted 2018-08-17 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Blood Pressure; Psychological Stress
Keywords: Non-Dipping Blood Pressure
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: All participants will be receive the same intervention.
Masking Description: All participants will receive the same intervention. All associated groups will be aware of the intervention protocol and the single-arm study model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychological Stress (Experimental): All enrolled participants who attended the laboratory visit underwent stress-inducing tasks (psychological stress) using validated research tools. Participants performed a 5-minute computer Stroop Color Test and a 5-minute verbal Mental Arithmetic Task. The research assistant asked the participant to work as quickly and accurately as possible for both tasks.
  Then during the ambulatory period, the participants underwent 24-hour ambulatory blood pressure monitoring during which urine was collected during the awake and asleep periods. Further, 5 ecological momentary assessment (EMA) ratings of perceived stress and negative affect (angry/hostile, aggravated/irritated, anxious/tense/nervous, and sad/blue/depressed) were collected during the awake period.
  Interventions: Behavioral: Psychological Stress Intervention

INTERVENTIONS:
Behavioral: Psychological Stress Intervention — All enrolled participants who attended the laboratory visit underwent stress-inducing tasks (psychological stress) using validated research tools. Participants performed a 5-minute computer Stroop Color Test and a 5-minute verbal Mental Arithmetic Task. The research assistant asked the participant to work as quickly and accurately as possible for both tasks.
  Other Names: Provoked Psychological Stress

SUMMARY:
The study will examine urinary sodium excretion induced by psychological stress and its diurnal pattern as a novel biological mechanism that may underlie an abnormal diurnal pattern of blood pressure. The study will test the hypotheses that lower stress-induced sodium excretion is associated with an abnormal diurnal pattern of sodium excretion, and that an abnormal diurnal pattern of sodium excretion is associated with an abnormal diurnal pattern of blood pressure.

Primary Aim 1: To examine the association between urinary sodium excretion after provoked psychological stress and the diurnal pattern of sodium excretion.

Primary Aim 2: To examine the association between the diurnal pattern of sodium excretion and the diurnal pattern of BP.

Secondary Aim: To examine whether the association between urinary sodium excretion after provoked stress and the diurnal pattern of sodium excretion is modified by ecological momentary levels of perceived stress, experienced during the daytime period.

Exploratory Aim: To determine the socio-demographic, behavioral, and psychological traits, chronic stress, and biological stress-related factors that are associated with lower stress-induced sodium excretion. Identification of these factors will help determine who is at risk for having a differential sodium excretion response to psychological stress.

DETAILED DESCRIPTION:
Blood pressure (BP) has a diurnal rhythm; it is normally highest during the daytime period and lowest during the nighttime period (BP dipping). The diurnal pattern of BP over a 24-hour period can be assessed using ambulatory BP monitoring (ABPM). Evidence indicates that an abnormal diurnal pattern of BP on ABPM, defined by reduced BP dipping or elevated nighttime BP, is associated with an increased risk of cardiovascular disease (CVD) events.

Psychological stress occurs when an individual perceives that the environmental demands exceed his/her adaptive capacity. An individual's response to events that are representative of this overload, such as perceived stress and negative affect including anger, hostility, depression, vital exhaustion, and symptoms of posttraumatic stress disorder, are associated with reduced BP dipping and/or higher nighttime BP. Exposure to environmental factors which tax an individual's ability to cope, including lower socioeconomic status, job strain, and perceived racism, are also associated with reduced BP dipping and/or higher nighttime BP. This study will examine the disruption of the normal diurnal pattern of sodium excretion by psychological stress as a novel biological mechanism underlying an abnormal diurnal pattern of BP.

The study will be conducted both in the laboratory and in the naturalistic environment with a multi-ethnic sample of 211 adult community participants from upper Manhattan who do not have a history of CVD, diabetes, chronic kidney disease, or another major medical condition and are not taking antihypertensive medication. During a laboratory visit, urinary sodium excretion in response to mental stress tasks will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* Screening mean blood pressure less than or equal to 160/105 mm Hg

Exclusion Criteria:

* History of overt cardiovascular disease (coronary heart disease, stroke, peripheral arterial disease, heart failure, permanent or recurring arrhythmia)
* History of secondary hypertension
* History of other major medical condition (cancer, rheumatologic diseases, immunologic diseases, etc.)
* Taking anti-hypertensive medications or other medications that are known to substantially affect blood pressure (e.g. steroids, chronic anti-inflammatory medications, etc.)
* Non-English speaking

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daichi Shimbo, MD, Principal Investigator — Professor of Medicine, Dept of Med Beh Cardiology
Locations (1):
- Columbia University Medical Center - Shimbo Hypertension Lab, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Psychological Stress: All enrolled participants who attended the laboratory visit underwent stress-inducing tasks (psychological stress) using validated research tools. Participants performed a 5-minute computer Stroop Color Test and a 5-minute verbal Mental Arithmetic Task. The research assistant asked the participant to work as quickly and accurately as possible for both tasks.
  Then the participants underwent 24-hour ambulatory blood pressure monitoring during which urine was collected during the awake and asleep periods. Further, 5 ecological momentary assessment (EMA) ratings of perceived stress and negative affect (angry/hostile, aggravated/irritated, anxious/tense/nervous, and sad/blue/depressed) were collected during the awake period.
Period: Overall Study
Arm/Group | Psychological Stress
Started | 323
Completed | 182
Not Completed | 141
Not completed — Dropped out or incomplete data | 141

BASELINE CHARACTERISTICS:
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.4 (10.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 113
  Male | 68
  Prefers not to identify | 1
  Unknown | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38
  Not Hispanic or Latino | 144
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 51
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 76
  More than one race | 25
  Unknown or Not Reported | 5
Current smoking [Count of Participants; unit: Participants]
  Yes | 5
  No | 177
Alcohol use [Count of Participants; unit: Participants]
  None | 71
  Moderate | 108
  Heavy | 3
Parental history of hypertension [Count of Participants; unit: Participants]
  Yes | 67
  No | 115
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 24.3 (4.6)
Systolic blood pressure (baseline) [Mean (Standard Deviation); unit: mm Hg] | 111.0 (10.5)
Diastolic blood pressure (baseline) [Mean (Standard Deviation); unit: mm Hg] | 72.2 (6.9)
Glucose [Mean (Standard Deviation); unit: mg/dL] | 89.1 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Awake-to-asleep Urinary Sodium Excretion Rate (Aim 1)
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: Ratio of awake-to-asleep
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
Ratio of awake-to-asleep | 1.4 (1.3)
Statistical Analysis 1: Comparison: Psychological Stress; Test type: Other — We tested an association between change in urinary sodium excretion rate with stress and ratio of awake-to-asleep urinary sodium excretion rate; p = 0.0032, Regression, Linear; Adjusted for age, sex, race, ethnicity, body mass index, mean DBP during the baseline period, and 24-hour creatinine clearance; unstandardized B coefficients = 0.0021, 95% CI [0.0007 to 0.0034]

2. Primary Outcome: Systolic Blood Pressure Dipping (Aim 2)
Description: Systolic blood pressure (SBP) dipping refers to the normal physiological decline in SBP during nighttime sleep. SBP dipping (%) was calculated as 100 * (mean awake SBP - mean asleep SBP) / (mean awake SBP).
Time Frame: Over 24-hour ambulatory period
Population: Of the 182 participants, 175 had complete data on ratio of awake-to-asleep urinary excretion rate and SBP dipping, and high-quality urine collection.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Psychological Stress
Number analyzed (Participants) | 175
percent | 14.3 (6.0)
Statistical Analysis 1: Comparison: Psychological Stress; Test type: Other — We tested an association between ratio of awake-to-asleep urinary sodium excretion rate and SBP dipping; p = 0.037, Regression, Linear; Adjusted for age, sex, race, ethnicity, BMI, smoking, alcohol use, glucose, 24-hr sodium and potassium excretion, 24-hr creat clear, and FENa; unstandardized B coefficients = 0.8244, 95% CI [0.0487 to 1.6000] — Data are unstandardized B coefficients (95% CI)

3. Secondary Outcome: Mean Perceived Stress Level
Description: This is to measure the ecological stress level for the awake period during which the participants' sodium excretion is monitored. A 10-point Visual Analog Scale (VAS) (0=Not at all, 5=Moderately, and 10=Extremely) was used to assess stress.
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
score on a scale | 1.5 (1.5)

4. Secondary Outcome: 24-hour Sodium Excretion
Description: Rate of sodium excretion, measured from urine collected from participants during the ambulatory period.
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: mmol/24 hours
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
mmol/24 hours | 121.8 (51.4)

5. Secondary Outcome: 24-hour Potassium Excretion
Description: Rate of potassium excretion, measured from urine collected from participants during the ambulatory period.
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: mmol/24 hours
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
mmol/24 hours | 53.7 (22.8)

6. Secondary Outcome: 24-hour Creatinine Clearance
Description: Rate of creatine clearance, measured from urine collected from participants during the ambulatory period.
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
mL/min | 112.7 (34.0)

7. Secondary Outcome: Fractional Excretion of Sodium
Description: Fractional excretion of sodium is the amount of sodium that leaves the body through urine compared to the amount filtered and reabsorbed by the kidney.
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
percent | 0.5 (0.2)

8. Secondary Outcome: EMA Stress
Description: 10-point Ecological Momentary Assessment (EMA) measures self-reported stress through a questionnaire (0=Not at all, 5=Moderately, and 10=Extremely). Higher score indicates worse stress. The average EMA score over 5 time points in a 24-hour ambulatory period are reported.
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
Score on a scale | 1.5 (1.5)

9. Secondary Outcome: EMA Anger
Description: 10-point Ecological Momentary Assessment (EMA) measures self-reported anger through a questionnaire (0=Not at all, 5=Moderately, and 10=Extremely). Higher score indicates worse anger. The average EMA score over 5 time points in a 24-hour ambulatory period are reported.
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
Score on a scale | 0.5 (1.1)

10. Secondary Outcome: EMA Aggravation
Description: 10-point Ecological Momentary Assessment (EMA) measures self-reported aggravation/irritation through a questionnaire (0=Not at all, 5=Moderately, and 10=Extremely). Higher score indicates worse aggravation. The average EMA score over 5 time points in a 24-hour ambulatory period are reported.
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
Score on a scale | 0.8 (1.2)

11. Secondary Outcome: EMA Anxiety
Description: 10-point Ecological Momentary Assessment (EMA) measures self-reported anxiety through a questionnaire (0=Not at all, 5=Moderately, and 10=Extremely). Higher score indicates worse anxiety. The average EMA score over 5 time points in a 24-hour ambulatory period are reported.
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
Score on a scale | 1.2 (1.4)

12. Secondary Outcome: EMA Depressed
Description: 10-point Ecological Momentary Assessment (EMA) measures self-reported sadness/depression through a questionnaire (0=Not at all, 5=Moderately, and 10=Extremely). Higher score indicates worse depression. The average EMA score over 5 time points in a 24-hour ambulatory period are reported.
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
Score on a scale | 0.6 (1.2)

13. Other Pre Specified Outcome: Change in Urinary Sodium Excretion Rate With Stress
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: uEq/min
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
uEq/min | 116.4 (125.4)

14. Other Pre Specified Outcome: Systolic Blood Pressure Dipping
Description: as for outcome 2
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
percent | 13.9 (6.5)

15. Other Pre Specified Outcome: Diastolic Blood Pressure Dipping
Description: Diastolic blood pressure (DBP) dipping refers to the normal physiological decline in DBP during nighttime sleep. DBP dipping (%) was calculated as 100 * (mean awake DBP - mean asleep DBP) / (mean awake DBP).
Time Frame: Over 24-hour ambulatory period
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Psychological Stress
Number analyzed (Participants) | 182
percent | 19.9 (7.9)

ADVERSE EVENTS:
Time Frame: For 3 days prior to the laboratory visit through the completion of the ambulatory period, up to 1 week.
Description: Adverse events were assessed by direct observation during the lab session, and self-report during the ambulatory session.
Arm/Group | Psychological Stress
All-Cause Mortality (participants affected / at risk) | 0/323
Serious Adverse Events (participants affected / at risk) | 0/323
Other Adverse Events (participants affected / at risk) | 0/323

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-01-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT03636490/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT03636490/SAP_001.pdf